CLINICAL TRIAL: NCT06657950
Title: Adaptation and Pilot Study of Integrative Yoga and Mindful Self-Compassion (I-YMSC) to Improve Mood in Women Survivors of Interpersonal Violence
Brief Title: Treatments for Improving Mood in Women Survivors of Interpersonal Violence: A Community-Engaged Study-1.2
Acronym: I-YMSC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2203-003 Open; K23AT011917 (NIH)
Record Dates: First submitted 2024-10-21; First posted 2024-10-26 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Distress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Integrative hatha yoga and mindful self-compassion (Experimental): 12 weeks of adapted, integrative yoga and mindful self-compassion specifically designed to be administered to women survivors of interpersonal violence.
  Interventions: Behavioral: Integrative hatha yoga and mindful self-compassion

INTERVENTIONS:
Behavioral: Integrative hatha yoga and mindful self-compassion — 12 weeks of integrative hatha yoga and mindful self-compassion training

SUMMARY:
Phase 1.2: Open Trial N=15 women survivors of interpersonal violence will be enrolled into a single-arm pilot trial to test the adapted integrative hatha yoga and mindful self-compassion program.

DETAILED DESCRIPTION:
In Phase 1.2, the investigators will conduct an open single-arm pilot trial of a 12 week adapted integrative hatha yoga and self-compassion program.

The investigators will enroll 15 women survivors of interpersonal violence in the open pilot trial.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Ages 18-65
3. Report having experienced interpersonal violence (defined to include all forms throughout the lifespan, confirmed with the Trauma History Questionnaire (THQ])
4. Report being distressed, defined by a score of >5 on the Kessler-6 screener
5. Speak and understand English well enough to understand questionnaires when they are read aloud
6. Have access to a telephone through owning one, a relative/friend, or an agency
7. Have access to a device that will support use of the video platform we are using to conduct assessments and for home practice yoga video sessions

Exclusion Criteria:

1. Inability to be physically active, determined by a score >1 on the Physical Activity Readiness Questionnaire (PAR-Q) and physician non-consent of participation
2. Planned surgery in next 6 months, as this would interfere with study participation
3. Pregnancy, as yoga should be modified for pregnancy

   Women who meet criteria for the following:
4. Current mania as determined by the Diagnostic Interview for Anxiety, Mood, and OCD and Related Neuropsychiatric Disorders (DIAMOND)
5. Lifetime history of psychotic disorders (DIAMOND)
6. Current probable severe substance use disorder (DIAMOND)
7. Current diagnosis of anorexia nervosa or history in past year (DIAMOND)
8. Moderate or high risk for suicide on the adapted Columbia Suicide Severity Rating Scale screen version-recent (C-SSRS) and/or endorsement of suicidal plan/intent in the past 3 months
9. Non-stable course of psychiatric treatments (medication, psychotherapy) for the last 8 weeks
10. Plan to move from the area in the next 6 months, as this may preclude study participation given enrollment timeframes
11. Self-report of experiencing intimate partner violence currently or within past six months (assessed by the Revised Conflict Tactics Scale 2 [R-CTS2]), as this would require a different type of intervention
12. Current weekly yoga practice or current participation in mindfulness-based programming, as these are the study interventions

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Feasibility | Post intervention (month 3)
  Feasibility assessed based on number of participants who remained in the intervention (retention).
Feasibility of Intervention Measure | Post intervention (month 3)
  The Feasibility of Intervention Measure (FIM) construct comprises four items with each item measured on a 1-5 scale. The total score range is from 4-20. Higher scores indicate greater feasibility.
Intervention Appropriateness Measure | Post intervention (month 3)
  The Intervention Appropriateness Measure (IAM) construct comprises four items with each item measured on a 1-5 scale. The total score range is from 4-20. Higher scores indicate greater feasibility.
Acceptability of Intervention Measure | Post intervention (month 3)
  The Acceptability of Intervention Measure (AIM) comprises four items with each item measured on a 1-5 scale. The total score range is from 4-20. Higher scores indicate greater feasibility.
The Client Satisfaction Questionnaire (CSQ-8) | Post intervention (month 3)
  Satisfaction with treatment assessed with The Client Satisfaction Questionnaire (CSQ-8). The CSQ-8 is an 8-item measure with each item measured on a 1-4 scale, and total score range from 8-32. Higher scores indicate greater client satisfaction.
Systematic Assessment of Treatment-emergent Events-general Inquiry (SAFTEE) | Mid intervention (month 1.5) and Post intervention (month 3)
  Participant safety/adverse events will be measured using the SAFTEE. Participants will also be asked weekly if they experienced any injuries as a result of yoga.

SECONDARY OUTCOMES:
Depression Anxiety and Stress Scale (DASS-21) | Post intervention (month 3)
  Distress at Month 3. The DASS-21 is a 21-item measure with each item measured on a 0-3 scale, and total score conversion ranging from 0-63. Higher global scores indicate greater psychological distress.

CONTACTS AND LOCATIONS:
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided